CLINICAL TRIAL: NCT06161337
Title: ChronoMet: Metabolic and Inflammatory Effects of Eating Timing and Quantity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MED-2023-32162
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Meals

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): 60 young (age 18-65), healthy, normal body mass index subjects for this study.
  Interventions: Dietary Supplement: Meals

INTERVENTIONS:
Dietary Supplement: Meals — Each subject will participate in 4 visits with a 1-week washout period in between visits.
  Each visit will be either a morning or evening consumption of either a standardized mixed meal of containing 600 calories (standard control) or 2400 calories (overeating meal) - meals will have the same nutrient composition.

SUMMARY:
This is an observational study to address the important knowledge gap of the metabolic and inflammatory impact of acute overeating and whether timing of acute overeating may modify these effects. The hypothesis is that acute overconsumption of calories will promote inflammation and metabolic dysfunction, with the most detrimental effects observed with evening caloric overconsumption. The expectation is that this study to provide critical insights into the biological consequences of overeating, which will direct novel approaches combating overeating and its detrimental health effects.

ELIGIBILITY:
Inclusion Criteria:

* ages of 18-65 years old
* not pregnant
* no comorbid conditions
* normal BMI (18.5 - 24.9 kg/m2)
* Weight ≥120 lbs self-reported weight

Exclusion Criteria:

* N/A

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2026-03-05 (Estimated); Study Completion 2027-03-05 (Estimated)

PRIMARY OUTCOMES:
Inflammatory markers quantification | 8 months
  employ a the MILLIPLEX ® Human Cytokine/Chemokine Multiplex Assay Panel to quantify 50 specific inflammatory markers in the serum samples.
quantitative metabolomics on serum samples | 8 months
  leverage the University of Minnesota Center for Metabolomics and Proteomics to conduct analysis of serum samples utilizing the Biocrates MxP Quant 500, which provides detailed quantification of over 500 individual metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Chow, MD,MS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States